CLINICAL TRIAL: NCT03308877
Title: Brief Intervention for Justice-Involved Substance Users: Moderators and Mechanisms of Change
Brief Title: Brief Intervention for Justice-Involved Substance Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc Swogger, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB69167; R01DA043660 (NIH)
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Substance Use; Violence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Motivational Intervention (BMI) (Experimental)
  Interventions: Behavioral: BMI; Behavioral: Stadard Care (SC)
- Standard Care (SC) (Active Comparator)
  Interventions: Behavioral: Stadard Care (SC)

INTERVENTIONS:
Behavioral: BMI — Four 45-minute, brief motivational sessions for substance use
  Arms: Brief Motivational Intervention (BMI)
Behavioral: Stadard Care (SC) — Standard procedures at pretrial program + assessement

SUMMARY:
This is a randomized clinical trial to study ways of helping justice-involved people change to more healthy behavior.

ELIGIBILITY:
Inclusion Criteria:

* In Monroe County Pretrial Services Program

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pretrial Services, Inc., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults were recruited from Pretrial Services subsequent to being charged with a crime. They were eligible for the trial if they had a Drug Abuse Screening Test (DAST) score at or above 3, indicating harmful substance use and provided informed consent to participate.
Period: Overall Study
Arm/Group | Brief Motivational Intervention (BMI) | Standard Care (SC)
Started | 70 | 62
6-week Assessment | 53 | 44
Completed (6-month (final) assessment) | 38 | 34
Not Completed | 32 | 28
Not completed — Lost to Follow-up | 32 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Motivational Intervention (BMI) | Standard Care (SC) | Total
Number analyzed (Participants) | 70 | 62 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 62 | 132
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.68 (11.70) | 36.06 (11.41) | 36.90 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 45 | 62
  Male | 53 | 17 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 23 | 18 | 41
  Race/Ethnicity: Black | 35 | 29 | 64
  Race/Ethnicity: Other | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 70 | 62 | 132
Timeline Followback; percent days abstinent [Mean (Standard Deviation); unit: percent days abstinent from alcohol/drug] | 34 (33) | 32 (40) | 33 (36)
Self-regulation Questionnaire [Mean (Standard Deviation); unit: units on a scale] — upper limit (high regulation) = 315; lower limit = 63
  units on a scale | 214.23 (25.07) | 211.37 (29.02) | 212.88 (26.94)
Alcohol use disorder identification test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — Upper limit (heavy drinking) = 40, lower limit = 0
  units on a scale | 14.23 (11.84) | 12.03 (11.53) | 13.19 (11.69)
Psychopathy Checklist Revised - total score [Mean (Standard Deviation); unit: units on a scale] — upper limit (high psychopathy)= 40, lower limit= 0
  units on a scale | 22.49 (7.15) | 21.14 (8.51) | 21.85 (7.79)
Readiness Ruler (readiness to change) [Mean (Standard Deviation); unit: units on a scale] — 1 (low readiness to change) to 10
  units on a scale | 6.71 (2.92) | 6.24 (2.78) | 6.49 (2.85)

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Abstinent
Description: Percent Days not using alcohol or drugs
Time Frame: 6 months
Population: Those who completed 6-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Brief Motivational Intervention (BMI) | Standard Care (SC)
Number analyzed (Participants) | 38 | 34
percentage of days abstinent | 44 (42) | 42 (41)
Statistical Analysis 1: Comparison: Brief Motivational Intervention (BMI) vs Standard Care (SC); Hypothesis 1: Affective psychopathy scores will moderate response to a BMI such that individuals with lower scores will benefit relative to controls, but individuals with higher psychopathy scores will not benefit from the intervention in terms of percent days abstinent; Test type: Other; p = .07, Regression, Linear — Covariates include education & percent days abstinent at baseline
Statistical Analysis 2: Comparison: Brief Motivational Intervention (BMI) vs Standard Care (SC); Sensitivity analysis: proximal follow-up (3 months following BMI or SC); Test type: Other; p = .02, Regression, Linear
Statistical Analysis 3: Comparison: Brief Motivational Intervention (BMI) vs Standard Care (SC); Increased readiness to change will be associated with decreased substance use; Test type: Other; p < .01, Regression, Linear; bias corrected bootstrap; B = .063, 95% CI 2-sided [.007 to .156]

2. Primary Outcome: Substance Use Consequences (SIP-AD)
Description: Short Inventory of Problems with Alcohol or Drugs (SIP-AD) Range 0-45 higher = more problems
Time Frame: 6 months
Population: Individuals who completed the 6-month follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Motivational Intervention (BMI) | Standard Care (SC)
Number analyzed (Participants) | 38 | 34
units on a scale | 14.55 (13.38) | 15.24 (13.79)
Statistical Analysis 1: Comparison: Brief Motivational Intervention (BMI) vs Standard Care (SC); Test type: Other; p = .74, Regression, Linear

3. Primary Outcome: Violent Charges
Description: Number of violent charges during follow-up from Statewide Database
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: violent charges during 2-year follow up
Arm/Group | Brief Motivational Intervention (BMI) | Standard Care (SC)
Number analyzed (Participants) | 36 | 28
violent charges during 2-year follow up | .48 (.97) | .43 (.92)
Statistical Analysis 1: Comparison: Brief Motivational Intervention (BMI) vs Standard Care (SC); Test type: Other; p = .88, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Brief Motivational Intervention (BMI) | Standard Care (SC)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/62
Other Adverse Events (participants affected / at risk) | 19/70 | 15/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Motivational Intervention (BMI) (N=70) | Standard Care (SC) (N=62)
Arrest; new criminal charges (Social circumstances) | 19 (19) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03308877/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03308877/SAP_001.pdf